CLINICAL TRIAL: NCT05308771
Title: Use of Visual Pressure Control (VPC) Syringes for Epidural Space Identification in Pediatric Anesthesia: a Pilot Study
Brief Title: To Investigate the Use of a New Syringe "Visual Pressure Control (VPC)" for Epidural Anesthesia in Children Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Tivoli (Other)
Responsible Party: Principal Investigator, Emmanuel Noel, Deputy head of anesthesiology department, Centre Hospitalier Universitaire de Tivoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VPC 1
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Abdominal Hernia; Abdominal Wall Defect; Abdominal Neoplasm; Urogenital Disease; Urologic Neoplasms; Thoracic Diseases; Lung Diseases
MeSH Terms: conditions — Hernia, Abdominal; Abdominal Neoplasms; Urogenital Diseases; Urologic Neoplasms; Thoracic Diseases; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Epidural anesthesia using VPC syringe (Experimental): Epidural anesthesia detection using VPC syringe
  Interventions: Device: VPC syringe

INTERVENTIONS:
Device: VPC syringe — Use of the visual pressure control syringe for epidural space detection

SUMMARY:
Pediatric epidural anesthesia has emerged as a safe and effective regional anesthesia technique for providing intraoperative and postoperative analgesia in thoracic and abdominal surgery. The loss of resistance technique is the gold standard for the placement of the epidural.

The VPC (visual pressure control) syringes developed by PAJUNK enable direct visualization of the introduction of the needle into the epidural space.

DETAILED DESCRIPTION:
This trial is a non blinded, pilot study. A minimum of 15 children between the ages of 0 and 16 who require surgery that may benefit from epidural anesthesia will be enrolled.

The number of attempts, the complications (dural and vascular punctures, neurological complications) and the degree of satisfaction of the operator measured by a 7-point likert scale will be studied as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 0 to 16y
* surgical procedure that can benefit from a lumbar or low thoracic epidural anesthesia

Exclusion Criteria:

* parental refusal
* allergy to local anesthetics
* coagulation disorders
* spine abnormalities

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
successful detection of the epidural space | 24 hours
  The primary objective will be successful detection of the epidural space by visualization of dural displacement upon injection of local anesthetic with real-time ultrasound and/or absence of pain at the incision established by the absence of more than 10% elevation in heart rate.

SECONDARY OUTCOMES:
Number of participants with vascular puncture | 24 hours
  puncture of a vessel with the epidural needle or catheter
Number of participants with dural puncture | 24 hours
  dura mater breach with needle
Number of participants with nerve damage | Month 3
  transient of permanent nerve damage
Operator's satisfaction questionnaire | 24 hours
  study of the operator's satisfaction by a seven-point rating scale where 1 is extremely dissatisfied and 7 is extremely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Noel, MD, Principal Investigator — Centre Hospitalier Universitaire de Tivoli
Locations (1):
- Chu Tivoli, La Louvière, Hainaut, Belgium

IPD SHARING:
Plan to Share IPD: No